CLINICAL TRIAL: NCT07337668
Title: The Effect of Mobile Application-Based Education Given to Patients With Tracheostomy on Depression, Social Adaptation and Quality of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Tracheostomy
Record Dates: First submitted 2026-01-04; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Tracheostomized Patients; Depression; Social Adaptation; Quality of Recovery
Keywords: mobile application; tracheostomy; education; quality of recovery; depression; social adaptation
MeSH Terms: conditions — Depression; Social Adjustment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this group received standard care plus a mobile application-based education program designed for patients with tracheostomy. The program included educational videos focusing on tracheostomy care, psychosocial support, and postoperative recovery.
  Interventions: Behavioral: Mobile application-based education
- Control group (Active Comparator): Participants in this group received standard postoperative care without access to the mobile application-based education program.
  Interventions: Other: Standart Care

INTERVENTIONS:
Behavioral: Mobile application-based education — A structured education program delivered via a mobile application for patients with tracheostomy. The program included educational videos focusing on tracheostomy care, and postoperative recovery. Participants accessed the content throughout the postoperative period in addition to standard care.
  Arms: Intervention group
Other: Standart Care — Standard postoperative care routinely provided to patients with tracheostomy according to institutional protocols
  Arms: Control group

SUMMARY:
The Effect of Mobile Application-Based Education Given to Patients with Tracheostomy on Depression, Social Adaptation and Quality of Recovery

DETAILED DESCRIPTION:
The Effect of Mobile Application-Based Education Given to Patients with Tracheostomy on Depression, Social Adaptation and Quality of Recovery

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Patients with a tracheostomy
* Able to communicate verbally or in writing
* Able to use a smartphone
* Provided written informed consent

Exclusion Criteria:

* Presence of severe cognitive impairment
* Presence of severe psychiatric disorder
* Patients with neurological diseases affecting swallowing
* Inability to use a mobile application
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-25 (Actual); Study Completion 2025-12-25 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline and postoperative 21 days
  Depression level was assessed using the Beck Depression Inventory
Social Adaptation | Baseline and postoperative 21 days
  Social adaptation was assessed using the Social Adaptation Self-evaluation Scale
Quality of Recovery | Postoperative 21 days
  Quality of recovery was assessed using the Quality of Recovery-40 (QoR-40) questionnaire.

SECONDARY OUTCOMES:
Swallowing Function | Baseline and postoperative 21 days
  Swallowing function was assessed using the Turkish version of the Eating Assessment Tool-10 (T-EAT-10).
Oral Care Status | Postoperative 21 days
  Oral care status was assessed using an oral care assessment too

CONTACTS AND LOCATIONS:
Locations (1):
- Basaksehir Cam and Sakura City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions and to protect participant confidentiality.

REFERENCES:
- [Background] Akkaya C, Sarandol A, Esen Danaci A, Sivrioglu EY, Kaya E, Kirli S. [Reliability and validity of the Turkish version of the Social Adaptation Self-Evaluation Scale (SASS)]. Turk Psikiyatri Derg. 2008 Fall;19(3):292-9. Turkish. PMID 18791882
- [Background] Demir N, Serel Arslan S, Inal O, Karaduman AA. Reliability and Validity of the Turkish Eating Assessment Tool (T-EAT-10). Dysphagia. 2016 Oct;31(5):644-9. doi: 10.1007/s00455-016-9723-9. Epub 2016 Jul 12. PMID 27405421
- [Background] Karaman S, Arici S, Dogru S, Karaman T, Tapar H, Kaya Z, Suren M, Gurler Balta M. Validation of the Turkish version of the Quality of Recovery-40 questionnaire. Health Qual Life Outcomes. 2014 Jan 15;12:8. doi: 10.1186/1477-7525-12-8. PMID 24428925
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369